CLINICAL TRIAL: NCT00318162
Title: Randomized Double-Blind Trial of Low-Dose Naltrexone for Children With PDD
Brief Title: Trial of Low-Dose Naltrexone for Children With Pervasive Developmental Disorder (PDD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Jerusalem Institute for Child Development (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PDDLDN-HMO-CTIL
Record Dates: First submitted 2006-04-25; First posted 2006-04-26 (Estimated); Last update posted 2006-05-03 (Estimated); Status verified 2006-04

CONDITIONS: Pervasive Developmental Disorder
Keywords: autism; PDD; LDN; naltrexone
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder | interventions — Naltrexone

INTERVENTIONS:
Drug: low dose naltrexone

SUMMARY:
This study will examine the effects of low-dose naltrexone (LDN) on children with autistic spectrum disorders. The investigators hope to show a positive effect on social functioning and language.

DETAILED DESCRIPTION:
Fifty children aged three to six years will be recruited for the study. They will be randomly assigned to receive either LDN or placebo for two months after which the treatment groups will be switched over. Assessments of functioning will be obtained from a video-taped play session, and by parent and teacher questionnaires at baseline, after two months and after four months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PDD

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)

PRIMARY OUTCOMES:
play observation
Autism Behavior Checklist (ABC) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David S Wilensky, MD, Principal Investigator — Jerusalem Institute for Child Development
Locations (1):
- Jerusalem Institute for Child Development, Jerusalem, Israel